CLINICAL TRIAL: NCT06357533
Title: A Phase III, Randomised, Open-label, Global Study of Datopotamab Deruxtecan (Dato-DXd) in Combination With Rilvegostomig or Rilvegostomig Monotherapy Versus Pembrolizumab Monotherapy for the First-line Treatment of Participants With Locally-advanced or Metastatic Non-squamous NSCLC With High PD-L1 Expression (TC ≥ 50%) and Without Actionable Genomic Alterations (TROPION-Lung10)
Brief Title: Phase III, Open-label, Study of First-line Dato-DXd in Combination With Rilvegostomig for Advanced Non-squamous NSCLC With High PD-L1 Expression (TC ≥ 50%) and Without Actionable Genomic Alterations
Acronym: TROPION-Lung10
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7632C00001; 2023-505077-32-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Non-Small Cell Lung Cancer; Datopotamab Deruxtecan; Rilvegostomig; Pembrolizumab; Non-squamous; PD-L1 expression >=50%; Locally-advanced NSCLC; Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Open-label, sponsor-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Datopotamab Deruxtecan in Combination With Rilvegostomig (Experimental): Participants in the Datopotamab Deruxtecan (Dato-DXd) in combination with Rilvegostomig group will receive Dato-DXd plus rilvegostomig as intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Interventions: Drug: Datopotamab Deruxtecan; Drug: Rilvegostomig
- Arm 2: Rilvegostomig Monotherapy (Experimental): Participants in the rilvegostomig monotherapy group will receive rilvegostomig as intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Interventions: Drug: Rilvegostomig
- Arm 3: Pembrolizumab Monotherapy (Active Comparator): Participants in the pembrolizumab group will receive pembrolizumab as intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Datopotamab Deruxtecan — Datopotamab Deruxtecan IV (intravenous)
  Other Names: Dato-DXd
  Arms: Arm 1: Datopotamab Deruxtecan in Combination With Rilvegostomig
Drug: Rilvegostomig — Rilvegostomig IV (intravenous)
  Other Names: AZD2936
  Arms: Arm 1: Datopotamab Deruxtecan in Combination With Rilvegostomig; Arm 2: Rilvegostomig Monotherapy
Drug: Pembrolizumab — Pembrolizumab IV (intravenous)
  Other Names: KEYTRUDA
  Arms: Arm 3: Pembrolizumab Monotherapy

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Dato-DXd in combination with rilvegostomig or rilvegostomig monotherapy compared with pembrolizumab monotherapy as a first line therapy in participants with locally advanced or metastatic non-squamous NSCLC with high PD-L1 expression (TC ≥ 50%) and without actionable genomic alterations.

DETAILED DESCRIPTION:
This is a Phase III, randomized, open-label, Global Study of Datopotamab Deruxtecan (Dato-DXd) in Combination With Rilvegostomig or Rilvegostomig monotherapy versus Pembrolizumab monotherapy for the first-line treatment of participants with locally-advanced or metastatic non-squamous NSCLC with high PD-L1 expression (TC ≥ 50%) and without actionable genomic alterations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented non-squamous NSCLC.
* Stage IIIB or IIIC or Stage IV metastatic NSCLC (according to Edition 8 of the AJCC staging manual) not amenable to curative surgery or definitive chemoradiation.
* Absence of sensitising EGFR mutations, and ALK and ROS1 rearrangements, and absence of documented local test result for any other known genomic alteration for which there are locally approved and available targeted first-line therapies.
* Must provide tumor sample to determine PD-L1 status, TROP2 status and other biomarkers.
* Known tumour PD-L1 expression status defined as TC ≥ 50%
* At least one lesion, not previously irradiated that qualifies as a RECIST 1.1 target lesion at baseline
* ECOG performance status of 0 or 1
* Adequate bone marrow reserve and organ function within 7 days before the first dose of study intervention

Exclusion Criteria:

* Prior systemic therapy for advanced/metastatic NSCLC.
* Squamous cell histology, or predominantly squamous cell histology NSCLC; mixed small cell lung cancer; NSCLC histology, sarcomatoid variant.
* History of another primary malignancy within 3 years
* Active or prior documented autoimmune or inflammatory disorders (with exceptions)
* Any evidence of severe or uncontrolled systemic diseases, including, but not limited to active bleeding diseases, active infection, active ILD/pneumonitis, cardiac disease.
* Has clinically significant third-space fluid retention (for example pleural effusion) and is not amenable for repeated drainage.
* History of non-infectious ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
* Has significant pulmonary function compromise, as determined by the investigator
* Spinal cord compression, or brain metastases unless participant treated and no longer symptomatic, radiologically stable, and who require no treatment with corticosteroids or anticonvulsants.
* History of leptomeningeal carcinomatosis
* Known clinically significant corneal disease
* Active infection with TB, HBV, HCV, Hepatitis A, or known HIV infection that is not well controlled
* History of active primary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2028-04-24 (Estimated); Study Completion 2030-05-24 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) in TROP2 biomarker positive participants. | Approximately 4 years
  PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause.
  The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy, receives another anti-cancer therapy or clinically progresses prior to RECIST 1.1 progression, in the following population:
  • TROP2 biomarker positive population
  The measure of interest is the HR of PFS. PFS by investigator will be reported as a sensitivity analysis.
Overall Survival (OS) in TROP2 biomarker positive participants. | Approximately 6 years
  OS is defined as the time from randomisation until the date of death due to any cause.
  The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anti-cancer therapy, in the following population:
  • TROP2 biomarker positive population The measure of interest is the HR of OS.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) in the FAS population. | Approximately 4 years
  PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause.
  The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy, receives another anti cancer therapy or clinically progresses prior to RECIST 1.1 progression, in the following population:
  • FAS population
  The measure of interest is the HR of PFS. PFS by investigator will be reported as a sensitivity analysis.
Overall Survival (OS) in the FAS population. | Approximately 6 years
  OS is defined as the time from randomisation until the date of death due to any cause.
  The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anti-cancer therapy, in the following population:
  • FAS population The measure of interest is the HR of OS.
Assessment of Objective Response Rate (ORR) by BICR in TROP2 biomarker positive and FAS populations | Approximately 4 years
  ORR is defined as the proportion of participants who have a CR or PR, as determined by BICR per RECIST 1.1.
  The analyses will include all randomised participants, as randomised, with measurable disease at baseline, in the following populations:
  * TROP2 biomarker positive population
  * FAS population Data obtained from randomisation up until progression, or the last evaluable assessment in the absence of progression, will be included in the assessment of ORR, regardless of whether the participant withdraws from therapy. Participants who go off treatment without a response or progression, receive a subsequent therapy, and then respond will not be included as responders in the ORR.
  The measure of interest is the OR of the ORR. ORR by investigator will be reported as a sensitivity analysis.
Assessment of Duration of Response (DoR) by BICR in TROP2 biomarker positive and FAS populations | Approximately 4 years
  DoR is defined as the time from the date of first documented response until date of documented progression per RECIST 1.1, as assessed by BICR and investigator assessment or death due to any cause.
  The analyses will include all randomised participants who have a response, as randomised, regardless of whether the participant withdraws from randomised therapy, receives another anti cancer therapy or clinically progresses prior to RECIST 1.1 progression, in the following populations:
  * TROP2 biomarker positive population
  * FAS population The measure of interest is the median of DoR. DoR by investigator will be reported as a sensitivity analysis.
Participant-reported lung cancer symptoms of NSCLC and participant-reported GHS/QOL in participants treated with Dato-DXd in combination with rilvegostomig relative to pembrolizumab. | Approximately 6 years
  Time to deterioration in: pulmonary symptoms (dyspnoea, cough, and chest pain) as measured by the NSCLC-SAQ, in overall lung cancer symptoms as measured by the NSCLC-SAQ, and in GHS/QoL as measured by the GHS/QoL scale from EORTC IL172.
  Time to deterioration is defined as the time from randomisation until the date of deterioration. Deterioration is defined as change from baseline that reaches a clinically meaningful deterioration threshold. The analyses will include all randomised participants, in the following populations:
  * TROP2 biomarker positive population
  * FAS population The measure of interest is the HR of time to deterioration in pulmonary symptoms, HR of time to deterioration in overall lung cancer symptoms, and HR of time to deterioration in GHS/QoL.
Participant-reported physical functioning in participants treated with Dato DXd in combination with rilvegostomig relative to pembrolizumab. | Approximately 6 years
  Time to deterioration in physical functioning as measured by PROMIS Physical Function short form 8c.
  Time to deterioration is defined as the time from randomisation until the date of deterioration. Deterioration is defined as change from baseline that reaches a clinically meaningful deterioration threshold. The analyses will include all randomised participants, in the following populations:
  * TROP2 biomarker positive population
  * FAS population The measure of interest is the HR of time to deterioration in physical functioning.
Pharmacokinetics (PK) | Approximately 6 years
  Concentration of rilvegostomig, Dato-DXd, total anti TROP2 antibody, and MAAA 1181a (payload deruxtecan) in plasma or serum and PK parameters (peak and trough concentrations).
Immunogenicity | Approximately 6 years
  Presence of ADA for Dato-DXd and rilvegostomig (confirmatory results, titres and neutralising antibodies for confirmed positive samples).
Second Progression-Free Survival (PFS2). | Approximately 6 years
  PFS2 is defined as the time from randomisation to the earliest of the progression events (following the initial progression), subsequent to first subsequent therapy, or death. Progression event includes radiological (RECIST 1.1) or clinical disease progression.
  The date of second progression will be recorded by the investigator in the eCRF and defined according to local standard practice.
  The analyses will include all randomised participants, as randomised, regardless of whether the participant withdraws from subsequent therapy and regardless of missed visits, in the following populations:
  * TROP2 biomarker positive population
  * FAS population The measure of interest is the HR of PFS2.

OTHER OUTCOMES:
Safety of Dato-DXd in combination with rilvegostomig and rilvegostomig monotherapy as compared with pembrolizumab. | Approximately 6 years
  Safety and tolerability will be evaluated in terms of AEs (graded by CTCAE Version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Suresh S. Ramalingam, MD, Principal Investigator — Emory University, Atlanta, Georgia, United States of America.
Locations (230):
- United States (52):
  - Research Site, Anchorage, Alaska
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Springdale, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Fountain Valley, California
  - Research Site, Newport Beach, California
  - Research Site, Clermont, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orange City, Florida
  - Research Site, Orlando, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Hinsdale, Illinois
  - Research Site, Noblesville, Indiana
  - Research Site, Annapolis, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Dearborn, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Hattiesburg, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Bozeman, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Stony Brook, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Perrysburg, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Greenville, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Odessa, Texas
  - Research Site, Fort Belvoir, Virginia
  - Research Site, Leesburg, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Vancouver, Washington
  - Research Site, Wenatchee, Washington
- Australia (8):
  - Research Site, Birtinya
  - Research Site, Blacktown
  - Research Site, Clayton
  - Research Site, Gosford
  - Research Site, Melbourne
  - Research Site, South Brisbane
  - Research Site, Southport
  - Research Site, Wodonga
- Austria (6):
  - Research Site, Innsbruck
  - Research Site, Krems
  - Research Site, Linz
  - Research Site, Rankweil
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (4):
  - Research Site, Anderlecht
  - Research Site, Hasselt
  - Research Site, La Louvière
  - Research Site, Liège
- Brazil (10):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Ipatinga
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, São Paulo
  - Research Site, Taubaté
- Canada (13):
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Rimouski, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Saskatoon, Saskatchewan
  - Research Site, Chicoutimi
- China (26):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Linhai
  - Research Site, Linyi
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- Germany (18):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Georgsmarienhütte
  - Research Site, Gera
  - Research Site, Gütersloh
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kempten
  - Research Site, Koblenz
  - Research Site, Ludwigsburg
  - Research Site, München
  - Research Site, Nuremberg
  - Research Site, Potsdam
  - Research Site, Ravensburg
- Hungary (10):
  - Research Site, Budapest
  - Research Site, Gyöngyös
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Salgótarján
  - Research Site, Szekszárd
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- India (9):
  - Research Site, Chennai
  - Research Site, Dwārka
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Marg Jaipur
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Thiruvananthapuram
- Italy (9):
  - Research Site, Bergamo
  - Research Site, Genoa
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Ravenna
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (23):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Hirosaki-shi
  - Research Site, Hiroshima
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kawasaki-shi
  - Research Site, Kumamoto
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Takaoka-shi
  - Research Site, Takatsuki-shi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Utsunomiya
  - Research Site, Yokohama
- Poland (4):
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Przemyśl
  - Research Site, Warsaw
- Research Site, San Juan, Puerto Rico
- South Korea (5):
  - Research Site, Changwon
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (5):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Jerez de la Frontera
  - Research Site, Reus,Tarragona
  - Research Site, Salamanca
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Muang
  - Research Site, Mueang
- Turkey (Türkiye) (5):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Diyarbakır
  - Research Site, Istanbul
- United Kingdom (5):
  - Research Site, Cheltenham
  - Research Site, Inverness
  - Research Site, London
  - Research Site, Preston
  - Research Site, Truro
- Vietnam (7):
  - Research Site, Da Nang
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Huế
  - Research Site, Vinh
  - Research Site, Vĩnh Yên

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.
  For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool .
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
  Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Newsom-Davis T, Melosky B, Heist RS, Lu S, Pasello G, Chen X, Stachowiak M, Lyfar P, Forcina A, Ramalingam SS. TROPION-Lung10: a phase 3 study of datopotamab deruxtecan and rilvegostomig in patients with treatment-naive locally advanced or metastatic nonsquamous non-small cell lung cancer with high PD-L1 expression and without actionable genomic alterations. Front Oncol. 2026 Jan 26;15:1721624. doi: 10.3389/fonc.2025.1721624. eCollection 2025. PMID 41669261